CLINICAL TRIAL: NCT03926247
Title: Addressing the Social-Structural Determinants of Mental Health Through Adaptation of a Transdisciplinary Ecological Intervention Model for Mexican Immigrants
Brief Title: Immigrant Well-being Project: Transdisciplinary Ecological Mental Health Intervention for Mexican Immigrants
Acronym: IWP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Jessica Goodkind, Associate Professor of Sociology, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22217; U54MD004811 (NIH)
Record Dates: First submitted 2019-04-12; First posted 2019-04-24 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Mental Health
Keywords: pilot study; mental health; immigrant; within-group longitudinal design
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a pilot study of an intervention with a within-group longitudinal design. All participants will participate in the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immigrant Well-being Project Intervention (Other): Intervention
  Interventions: Behavioral: Immigrant Well-Being Project

INTERVENTIONS:
Behavioral: Immigrant Well-Being Project — The IWP intervention emphasizes a sustainable and replicable partnership model between community-based organizations and universities that involves Mexican immigrants and undergraduate advocates working together to: a) increase immigrants' abilities to navigate their communities; b) improve immigrants' access to community resources; c) enhance meaningful social roles by valuing immigrants' culture, experiences, and knowledge; d) reduce immigrants' social isolation; and e) increase communities' responsiveness to immigrants through changes in policy and practice. The IWP is administered by university students enrolled in a service learning course, and has two elements: 1) Learning Circles, which involve cultural exchange and one-on-one learning opportunities, and; 2) Advocacy, which involves collaborative efforts to mobilize community resources related to health, housing, employment, education, and legal issues.

SUMMARY:
The goal of this study is to test a transdisciplinary ecological approach to reducing mental health disparities among Mexican immigrants by adapting and integrating a multilevel community-based advocacy, learning, and social support intervention (Immigrant Well-being Project, IWP) into existing efforts at three community partner organizations that focus on mental health, education, legal, and civil rights issues for Mexican immigrants. This research is innovative and significant because it employs cutting edge strategies to address social-structural determinants of mental health and examines the community-engaged process of adapting and testing the impact of a multilevel intervention originally designed for refugees. The IWP intervention emphasizes a sustainable and replicable partnership model between community-based organizations and universities that involves Mexican immigrants and undergraduate advocates working together to: a) increase immigrants' abilities to navigate their communities; b) improve immigrants' access to community resources; c) enhance meaningful social roles by valuing immigrants' culture, experiences, and knowledge; d) reduce immigrants' social isolation; and e) increase communities' responsiveness to immigrants through changes in policy and practice. The IWP is administered by university students enrolled in a service learning course, and has two elements: 1) Learning Circles, which involve cultural exchange and one-on-one learning opportunities, and; 2) Advocacy, which involves collaborative efforts to mobilize community resources related to health, housing, employment, education, and legal issues. Studies of the intervention model with refugees demonstrated feasibility, appropriateness, acceptability, and evidence that the intervention decreased participants' psychological distress and increased protective factors, and impacted changes in system-wide policies and practices. After completing in-depth ethnographic interviews with 24 Mexican immigrant adults to elucidate their mental health needs, stressors, current political/economic/social context, and local solutions, and a process of community engagement and intervention adaptation, a mixed methods strategy with data collected from 90 participants at four time points over a period of 14 months will be used to test the impact of the 6-month intervention on reducing psychological distress, increasing protective factors (access to resources, English proficiency, environmental mastery, and social support), and achieving system-level changes in organizational, local, and state policies and practices that impact Mexican immigrants' well-being. Mechanisms of intervention effectiveness will be explored by testing mediating relationships between protective factors and psychological distress. Qualitative data will explore feasibility and acceptability of the intervention, participants' experiences in the intervention, and unexpected impacts; document multilevel changes and the context of implementation at each site; and inform interpretation of quantitative data. Quantitative and qualitative data on the quality of the CBPR partnerships and their relationship to multilevel outcomes will also be examined.

DETAILED DESCRIPTION:
The goal of this research is to advance the science of community-level mental health interventions that aim to reduce social inequities and health disparities. The proposed study will adapt and integrate a successfully implemented multilevel, ecological intervention that addresses social-structural determinants of mental health into existing efforts at three community partner organizations that focus on mental health, education, legal, and civil rights issues for Mexican immigrants in New Mexico. Using a mixed methods longitudinal design, the processes and outcomes of the collaborative, community-based intervention efforts, including the impact of the quality of the community-based participatory research (CBPR) partnerships on individual, organizational, and community-level outcomes, will be illuminated.

Social and structural inequities contribute significantly to increasing health disparities globally, with the increasing numbers of migrants throughout the world bearing a disproportionate burden. The immigrant share of the U.S. population has risen steadily over the past four decades, comprising 13.5% of the total population in 2015, with Mexican-born immigrants accounting for 27% of all immigrants. The social, legal, and economic context of the migration process, including increasing uncertainty, discrimination, stigma, lack of access to resources, and fear of deportation and family separation based on immigration policies and public perception of immigrants as a threat all have a critical impact on adverse mental health outcomes among Mexican immigrants in the U.S. In addition, Mexican immigrants have low utilization rates for mental healthcare, in part because of barriers that include lack of health insurance, ineligibility for governmental health programs, discrimination, lack of interpretation services and culturally appropriate care, and an anti-immigrant political and economic climate. Although evidence points to the need to address socio-structural determinants, many mental health interventions offered to Mexican immigrants have focused on individual-level predictors of mental health. Also, Mexican immigrants' health outcomes are often viewed within the Latino health paradox, and therefore are frequently overlooked in mental health research and development of appropriate interventions, despite mounting evidence of mental health disparities and disproportionate exposure to trauma. Thus, multilevel, transdisciplinary intervention approaches that address social-structural determinants of mental health, are culturally appropriate, build upon Mexican immigrants' strengths, are cost-effective and scalable, and occur in non-stigmatized settings are needed.

In prior NIH-funded research, the PI and community partners developed and tested a 6-month community-based advocacy, learning, and social support intervention, which pairs paraprofessional university students with refugee adults to engage in mutual learning and social change efforts. The intervention was found to decrease participants' psychological distress, improve their quality of life, access to resources, social support, and English proficiency, and improve communities' responsiveness to refugees; and also proved to be highly acceptable, cost effective, and sustainable. The objective of this study is to: a) adapt the intervention for Mexican immigrants (Immigrant Wellbeing Project; IWP); b) integrate IWP into existing efforts at three community partner organizations; and c) elucidate new understandings of partnership and intervention processes that lead to sustainable multilevel changes and the reduction of mental health disparities and related social inequities.

Aim 1. Conduct an in-depth study of the mental health needs, stressors, current political/economic/social context, and local solutions as experienced by 24 Mexican recent and non-recent immigrants and their families residing in Bernalillo County New Mexico and contextualized by staff at three community partner organizations.

Aim 2. Building on the data from Aim 1, use a CBPR approach to adapt the intervention model (IWP) and integrate it within existing service delivery and social change efforts at three community partner organizations.

Aim 3. Using a mixed methods longitudinal design, investigate the feasibility and acceptability of the adapted community-based mental health intervention and test the quality of the CBPR partnership and impact of the intervention on mental health problems and protective factors among 90 Mexican immigrants and on organizational and government changes in policies and practices impacting immigrant mental health.

3.1 The IWP and collaborative adaptation/integration process will be feasible and acceptable and will serve as a model for implementing and studying multilevel, community-based intervention efforts.

3.2 IWP participants' psychological distress will decrease significantly over time.

3.3 IWP participants' protective factors (access to resources, English proficiency, environmental mastery, social support) will increase significantly over time.

3.4 Lower levels of psychological distress will be mediated by the protective factors.

3.5 Qualitative data will document changes in organizational and governmental policies and practices and the context of implementation at each site, explore other impacts, and inform interpretation of quantitative data.

3.6 Quality of CBPR partnership at each site will be related to policy/practice changes and health outcomes.

As one of the core research projects of the Transdisciplinary Research, Equity and Engagement Center for Advancing Behavioral Health (TREE), this study will benefit from and contribute to collaborative efforts to elucidate and address the impact of social-structural (e.g., racism, lack of access to resources) and historical (e.g., violence, trauma, colonization) determinants of mental health for immigrant and indigenous populations.

ELIGIBILITY:
Inclusion Criteria:

* Mexican immigrant
* Residing in Bernalillo County, New Mexico

Exclusion Criteria:

* Severe cognitive functioning problems
* Imminent suicide risk
* Mental illness that is so severe as to impede participation in a group and that warrants immediate individual treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica R Goodkind, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immigrant Well-being Project Intervention
Started | 56
Completed | 31
Not Completed | 25

BASELINE CHARACTERISTICS:
Population: A total of 56 participants enrolled in the study and completed the intervention. However, 2 of the participants did not complete the baseline interview (but completed interviews at subsequent time points).
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.06 (9.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 54
Region of Enrollment [Number; unit: participants]
  United States | 54
Perceived English Proficiency [Mean (Standard Deviation); unit: units on a scale] — Perceived English proficiency (Rumbaut, 1989) was measured as the mean of four items that asked participants to rate how well they understand, speak, read, and write English. Response choices ranged from 0 (not at all) to 3 (like a native), and total scores were calculated and averaged. Higher scores reflect higher degrees of perceived English proficiency.
  units on a scale | 1.12 (0.72)
Satisfaction with Resources [Mean (Standard Deviation); unit: units on a scale] — The Satisfaction with Resources Scale (Sullivan, et al., 1992) asks respondents to rate how satisfied they are with the resources they have in 11 specific domains (e.g., education, health care, housing, employment). Items are rated on a 7-point scale and averaged, with domain-specific scores ranging from 1 to 7. Higher scores reflect higher levels of perceived satisfaction with resources in the community
  units on a scale | 3.18 (1.00)
Difficulty Accessing Resources [Mean (Standard Deviation); unit: units on a scale] — The Difficulty Obtaining Resources scale (Sullivan & Bybee, 1999) asks participants to rate, on a 4-point scale, how difficult it had been or would be in the future to obtain resources they needed in the 12 specific life domains. Difficulty accessing resources was computed as the mean difficulty over all the resources respondents reported accessing (range 1 to 4); if they were not accessing a resource, their response was taken as their rating of how difficult they thought accessing that resource would be in the future. A higher score indicates more difficulty accessing resources.
  units on a scale | 2.51 (1.29)
Multisectoral Social Support Inventory [Mean (Standard Deviation); unit: units on a scale] — The Multi-Sector Social Support Inventory Scale (Layne et al., 2009) was used to assess perceived past-month social support in three domains: family, ethnic community, and nonethnic community. Each of the three parallel scales includes the same nine items related to subjective attachment and perceived support. Response choices range from 0 (never) to 4 (almost always), and total scores can range from 0 to 4. Higher scores indicate higher levels of social support.
  units on a scale | 2.14 (0.76)
Collective Efficacy [Mean (Standard Deviation); unit: units on a scale] — The Collective Efficacy Scale (Sampson et al., 1993) measures an individual's perception of how well communities collaborate to accomplish goals. This 10-item measure asks participants the likleihood of community action across scenarios from 1 (very likely) to 5 (very unlikely). Items are added and averaged, with lower scores indicating greater collective efficacy.
  units on a scale | 2.85 (0.88)
Social Cohesion [Mean (Standard Deviation); unit: units on a scale] — The Social Cohesion Scale (Li et al., 2015) is a five-item measure which assesses individual peception of community camraderie and belonging. Likert-type item responses range from 1 (strongly agree) to 4 (strongly disagree) with lower scores indicating stronger perception of social cohesion.
  units on a scale | 3.12 (0.85)
WHO Psychological Wellbeing [Mean (Standard Deviation); unit: units on a scale] — Three items (life enjoyment, life meaningfulness, and ability to concentrate) from the Psychological subscale of the World Health Organization Quality of Life Assessment (WHOQOL Group, 1998) were used to examine Psychological quality of life. Items are rated on a 5-point scale ranging from 1 (not at all) to 5 (an extreme amount) and summed for a subscale score with possible range of 3.00 to 15.00. Higher scores indicate higher perceived psychological quality of life.
  units on a scale | 10.51 (2.44)
WHO Physical Wellbeing [Mean (Standard Deviation); unit: units on a scale] — Three items (pain, need for medical treatment, energy) from the Physical subscale of the World Health Organization Quality of Life Assessment (WHOQOL Group, 1998) were used to examine physical quality of life. Items are rated on a 5-point scale ranging from 1 (not at all) to 5 (an extreme amount) and summed for a subscale score with possible range of 3.00 to 15.00. Higher scores indicate higher perceived physical quality of life.
  units on a scale | 8.60 (2.75)
WHO Environmental Wellbeing [Mean (Standard Deviation); unit: units on a scale] — Four items (safety, health of physical environment, access to needed information, opportunity for leisure activities) from the Environmental subscale of the World Health Organization Quality of Life Assessment (WHOQOL Group, 1998) were used to examine environmental quality of life. Items are rated on a 5-point scale ranging from 1 (not at all) to 5 (an extreme amount) and summed for a subscale score with possible range of 4.00 to 20.00. Higher scores indicate higher perceived environmental quality of life.
  units on a scale | 10.21 (2.87)
Hispanic Stress Inventory [Mean (Standard Deviation); unit: units on a scale] — The Hispanic Stress Inventory (Cervantes et al., 2015) is a measure of stress exposure to commonly experienced stressors for Hispanic communities. Responses range from 1 (Not at all worried/tense) to 5 (Extremely worried/tense) and are summed and averaged to develop a final score. A higher score indicates more stress.
  units on a scale | 1.31 (0.59)
Hopkins Symptom Checklist [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Symptom Checklist (HSC-25; Derogatis, 1974) is a self-report measure of anxiety and depressive symptoms that has been shown to be a valid measure of symptoms in refugee populations (Hollifield et al., 2002). Respondents rate 25 items on a Likert-type scale ranging from 1 (not at all) to 4 (extremely). Mean scores for items related to depression (15 items) and anxiety (10 items) can be calculated to create separate subscale scores (range: 1-4), with higher scores indicating higher levels of emotional distress.
  units on a scale | 1.61 (0.48)
HSC Depression Subscale [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Symptom Checklist (HSC-25; Derogatis, 1974) is a self-report measure of anxiety and depressive symptoms that has been shown to be a valid measure of symptoms in refugee populations (Hollifield et al., 2002). Respondents rate 25 items on a Likert-type scale ranging from 1 (not at all) to 4 (extremely). Mean scores for items related to depression (15 items) are calculated to create a separate depression subscale (range: 1-4), with higher scores indicating higher levels of depression symptoms.
  units on a scale | 1.64 (0.49)
HSC Anxiety Subscale [Mean (Standard Deviation); unit: units on a scale] — The Hopkins Symptom Checklist (HSC-25; Derogatis, 1974) is a self-report measure of anxiety and depressive symptoms that has been shown to be a valid measure of symptoms in refugee populations (Hollifield et al., 2002). Respondents rate 25 items on a Likert-type scale ranging from 1 (not at all) to 4 (extremely). Mean scores for items related to anxiety (10 items) are calculated to create a separate anxiety subscale (range: 1-4), with higher scores indicating higher levels of anxiety symptoms.
  units on a scale | 1.57 (0.51)
PTSD Symptom Checklist [Mean (Standard Deviation); unit: units on a scale] — The PTSD Symptom Checklist-Civilian Version (PCL-C; Weathers et al., 1993) is a 17-item self-reported measure of PTSD symptoms, per the criteria in the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Respondents rate answers on a scale ranging from 1 (not at all) to 5 (extremely). A total score is calculated (range: 17-85), with higher scores indicating higher PTSD symptom levels.
  units on a scale | 28.44 (12.35)
Trauma Exposure [Mean (Standard Deviation); unit: units on a scale] — Trauma exposure was assessed using a checklist with items from the Adolescent Self-Report Trauma Questionnaire (Horowitz et al., 1995), the Harvard Trauma Questionnaire (Mollica et al., 1992), and the PTSD Symptom Scale (Falsetti et al., 1993). A panel of researchers and cultural experts selected items for this study to best capture the experiences of these forcibly displaced groups. The checklist included 27 dichotomous items (1 for "yes," 0 for "no"), with scores ranging from 0 to 27. Higher scores indicate exposure to more traumatic events.
  units on a scale | 6.42 (5.26)
Resilience (CDRISC) [Mean (Standard Deviation); unit: units on a scale] — The Connor-Davidson Resilience scale (Connor & Davidson, 2003) is a measure of psychological resilience. Twenty-five items are rated on a 5-point scale (0-4), with higher scores reflecting greater resilience. For a final score, item responses are averaged.
  units on a scale | 2.70 (0.87)
Major Discrimination Scale [Mean (Standard Deviation); unit: units on a scale] — The 9-item Experiences of Discrimination instrument asks respondents whether they have ever experienced racial/ethnic discrimination in 9 different domains (involving work, school, housing, finances, medical care, service, public settings, and the police and courts). Two additional questions were included including legal status and speaking English. Response options are recorded dichotomously (0 = No; 1 = Yes) Items were combined and totaled with scores ranging from 0 to 11. Higher scores indicate more experiences of discrimination.
  units on a scale | 0.20 (0.18)
Everyday Discrimination Scale [Mean (Standard Deviation); unit: units on a scale] — The nine-item EDS (Williams et al. 1997) measures chronic and routine unfair treatment in everyday life. Adopted from the Detroit Area Study, respondents were asked to report how often they experience unfair treatment in their day-to-day life on a 6-point Likert-type response format. Response categories ranged from 0 (never) to 3 (four or more times), with higher scores indicating greater perceived everyday discrimination. Scores were summed and averaged. Scores can range from 0.00 to 3.00.
  units on a scale | 0.78 (0.64)
Work Discrimination Scale [Mean (Standard Deviation); unit: units on a scale] — The Work Discrimination and Harassment Scale (abbreviated) (Sternthall et al., 2011) is a six-item measure of experiences of discrimination in a workplace setting over a 12-month period. Responses to these items range from 1 (once a week or more) to 5 (never). Scores are summed and average, with lower final scores indicating higher experiences of workplace discrimination and harassment.
  units on a scale | 2.66 (1.65)
Heightened Vigilance Scale [Mean (Standard Deviation); unit: units on a scale] — The Heightened Vigilance Scale (abbreviated) (Hicken et al., 2016) is a four-item measure which assesses hypervigilance around one's perception by others, including how they might react negatively to ones dress, speech, and actions. Responses are reported on a scale of one (Almost every day) to 6 (Never), where lower scores indicate more hypervigilance around these issues. Items are averaged to total a final score.
  units on a scale | 2.96 (1.03)

OUTCOME MEASURES:

1. Primary Outcome: Linear Change From Baseline to 14-month Follow-up in Depression/Anxiety Symptom Score Assessed by the Hopkins Symptom Checklist-25
Description: Hopkins Symptom Checklist-25 (HSC-25). Minimum=1.00, Maximum=4.00. Lower scores indicate better outcome (lower levels of depression/anxiety symptoms).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: 56 participants enrolled in the study and participated in the intervention; we included participants in a particular outcome analysis if they had data for the outcome at a minimum of two timepoints (one of which had to be either the first or second timepoint).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 39
score on a scale
  Timepoint 1 (Baseline): number analyzed (Participants) | 37
  Timepoint 1 (Baseline) | 1.60 (0.08)
  Timepoint 2 (Mid-Intervention): number analyzed (Participants) | 38
  Timepoint 2 (Mid-Intervention) | 1.56 (0.07)
  Timepoint 3 (Post-Intervention): number analyzed (Participants) | 33
  Timepoint 3 (Post-Intervention) | 1.47 (0.08)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 36
  Timepoint 4 (8-month follow-up) | 1.49 (0.08)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' depression/anxiety symptoms would decrease overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups); p = 0.019, Mixed Models Analysis; LSM Final Difference = -0.044, 95% CI 2-sided [-0.087 to -0.008], Standard Error of Mean 0.019

2. Primary Outcome: Linear Change From Baseline to 14-month Follow-up in PTSD Symptom Score Assessed by the PTSD Symptom Checklist (Civilian Version)
Description: PTSD Symptom Checklist (Civilian Version, PCL-C). Minimum=17.00, Maximum=85.00. Lower scores indicate better outcome (lower levels of PTSD symptoms).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 38
score on a scale
  Timepoint 1 (Pre-intervention): number analyzed (Participants) | 37
  Timepoint 1 (Pre-intervention) | 28.72 (1.99)
  Timepoint 2 (Mid-intervention) | 29.34 (1.99)
  Timepoint 3 (Post-intervention): number analyzed (Participants) | 33
  Timepoint 3 (Post-intervention) | 25.32 (2.05)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 36
  Timepoint 4 (8-month follow-up) | 27.05 (2.00)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' PTSD symptoms would decrease overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups); p = 0.168, Mixed Models Analysis; Mean Difference (Final Values) = -0.892, 95% CI 2-sided [-2.161 to 0.372], Standard Error of Mean 0.643

3. Primary Outcome: Linear Change From Baseline to 14-month Follow-up in Stress Assessed by the Abbreviated Hispanic Stress Inventory Scale - Culturally-Specific Distress
Description: Abbreviated Hispanic Stress Inventory. Minimum=0.00, Maximum=3.00. Lower scores indicate better outcome (lower levels of stress). We adapted this measure for our study - based on community member input, we reduced response choices to 4 (from 5).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 32
score on a scale
  Timepoint 1 (Baseline) | 1.32 (0.11)
  Timepoint 2 (Mid-intervention): number analyzed (Participants) | 28
  Timepoint 2 (Mid-intervention) | 1.38 (0.11)
  Timepoint 3 (Post-intervention): number analyzed (Participants) | 28
  Timepoint 3 (Post-intervention) | 1.16 (0.11)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 28
  Timepoint 4 (8-month follow-up) | 1.18 (0.12)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' stress would decrease overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups); p = 0.051, Mixed Models Analysis; Mean Difference (Final Values) = -0.061, 95% CI 2-sided [-0.140 to -0.000], Standard Error of Mean 0.035

4. Secondary Outcome: Linear Change From Baseline to 14-month Follow-up in Social Support Assessed by the Multi-Sector Social Support Inventory
Description: Multi-Sector Social Support Inventory. Minimum=0.00, Maximum=4.00. Higher scores indicate better outcome (higher levels of social support).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 39
score on a scale
  Timepoint 1 (Baseline): number analyzed (Participants) | 37
  Timepoint 1 (Baseline) | 2.32 (0.11)
  Timepoint 2 (Mid-intervention): number analyzed (Participants) | 38
  Timepoint 2 (Mid-intervention) | 2.32 (0.11)
  Timepoint 3 (Post-intervention): number analyzed (Participants) | 33
  Timepoint 3 (Post-intervention) | 2.29 (0.12)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 36
  Timepoint 4 (8-month follow-up) | 2.21 (0.12)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' social support would increase overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups); p = 0.211, Mixed Models Analysis; Mean Difference (Final Values) = -0.041, 95% CI 2-sided [-0.106 to 0.023], Standard Error of Mean 0.029

5. Secondary Outcome: Linear Change From Baseline to 14-month Follow-up in Access to Resources Assessed by the Satisfaction With Resources Scale
Description: Satisfaction with Resources Scale. Minimum=0.00, Maximum=6.00. Higher scores indicate better outcome (higher satisfaction with resources).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 28
score on a scale
  Timepoint 1 (Baseline): number analyzed (Participants) | 24
  Timepoint 1 (Baseline) | 3.15 (0.18)
  Timepoint 2 (Mid-intervention) | 3.46 (0.17)
  Timepoint 3 (Post-intervention): number analyzed (Participants) | 20
  Timepoint 3 (Post-intervention) | 3.55 (0.18)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 26
  Timepoint 4 (8-month follow-up) | 3.43 (0.17)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' access to resources would increase overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups); p = 0.074, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.008 to 0.201], Standard Error of Mean 0.053

6. Secondary Outcome: Linear Change From Baseline to 14-month Follow-up in Access to Resources Assessed by the Difficulty Accessing Resources Scale
Description: Difficulty Accessing Resources Scale. Minimum=1.00, Maximum=4.00. Lower scores indicate better outcome (lower levels of difficulty accessing resources).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 34
score on a scale
  Timepoint 1 (Baseline): number analyzed (Participants) | 32
  Timepoint 1 (Baseline) | 2.55 (0.15)
  Timepoint 2 (Mid-intervention): number analyzed (Participants) | 32
  Timepoint 2 (Mid-intervention) | 2.34 (0.15)
  Timepoint 3 (Post-intervention): number analyzed (Participants) | 26
  Timepoint 3 (Post-intervention) | 2.46 (0.17)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 31
  Timepoint 4 (8-month follow-up) | 2.16 (0.15)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' difficulty accessing resources would decrease overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups)=; p = 0.089, Mixed Models Analysis; Mean Difference (Final Values) = -0.119, 95% CI 2-sided [-0.257 to 0.017], Standard Error of Mean 0.061

7. Secondary Outcome: Linear Change From Baseline to 14-month Follow-up in Quality of Life Assessed by the World Health Organization Quality of Life Assessment
Description: World Health Organization Quality of Life assessment (WHOQOL). Minimum=3.00, Maximum=15.00. Higher scores indicate better outcome (higher quality of life).
Time Frame: Timepoints used in calculation: baseline, 3 months (mid), 6 months (post), 14 months (follow-up)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Immigrant Well-being Project Intervention
Number analyzed (Participants) | 39
units on a scale
  Timepoint 1 (Baseline): number analyzed (Participants) | 37
  Timepoint 1 (Baseline) | 10.40 (0.38)
  Timepoint 2 (Mid-intervention): number analyzed (Participants) | 38
  Timepoint 2 (Mid-intervention) | 10.55 (0.38)
  Timepoint 3 (Post-intervention): number analyzed (Participants) | 32
  Timepoint 3 (Post-intervention) | 10.68 (0.40)
  Timepoint 4 (8-month follow-up): number analyzed (Participants) | 36
  Timepoint 4 (8-month follow-up) | 9.73 (0.38)
Statistical Analysis 1: Comparison: Immigrant Well-being Project Intervention; Analyses were conducted using a mixed effects linear model to calculate least square means across the 4 timepoints. This was a longitudinal within-group analysis with 4 timepoints of data nested within 56 individuals. Our hypothesis was that participants' quality of life would increase overtime; Test type: Other — Within-group longitudinal analysis (no comparison groups); p = 0.086, Mixed Models Analysis; Mean Difference (Final Values) = -0.216, 95% CI 2-sided [-0.461 to 0.030], Standard Error of Mean 0.124

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Immigrant Well-being Project Intervention
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT03926247/Prot_SAP_000.pdf